CLINICAL TRIAL: NCT00487084
Title: Interaction Between Epidural 2-chloroprocaine and Epidural Morphine: Effect of Timing on Efficacy of Morphine Analgesia After 2-chloroprocaine Anesthesia
Brief Title: Effect of Timing on Efficacy of Morphine Analgesia After 2-chloroprocaine Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Cynthia Wong, Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524-021
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Results first posted 2011-04-18 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Labor; Analgesia, Epidural
Keywords: analgesia; tubal ligation; chloroprocaine
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- morphine - 2CP-saline (MCS) (Experimental): morphine will be administered 30 min prior to epidural anesthesia; 2CP will be used to achieve a T4 level; saline will be administered at skin incision
  Interventions: Drug: Morphine-CP-saline (MCS)
- saline-2CP-morphine (SCM) (Experimental): saline will be administered 30 min prior to epidural anesthesia; 2CP will be used to achieve a T4 level;morphine will be administered at skin incision
  Interventions: Drug: saline-2CP-morphine (SCM)
- saline-lidocaine-morphine (SLM) (Active Comparator): Saline will be administered 30 min prior to epidural anesthesia; lidocaine will be used to achieve a T4 level; morphine will be administered at skin incision
  Interventions: Drug: saline-lidocaine-morphine (SLM)

INTERVENTIONS:
Drug: Morphine-CP-saline (MCS) — 3mg of preservative free morphine will be administered epidurally 30 min prior to epidural anesthesia. Epidural 3% 2CP will be used to achieve a T4 dermatomal level for surgical anesthesia for PPTL. 6ml of epidural saline will be administered at skin incision
  Arms: morphine - 2CP-saline (MCS)
Drug: saline-2CP-morphine (SCM) — 6ml of saline will be administered epidurally 30 min prior to epidural anesthesia. Epidural 3% 2CP will be used to achieve a T4 dermatomal level for surgical anesthesia for PPTL. 3mg of preservative free morphine will be administered at skin incision
  Arms: saline-2CP-morphine (SCM)
Drug: saline-lidocaine-morphine (SLM) — 3mg of preservative free morphine will be administered epidurally 30 min prior to epidural anesthesia. Epidural 2% lidocaine with epinephrine 1:200,000 will be used to achieve a T4 dermatomal level for surgical anesthesia for PPTL. 6ml of epidural saline will be administered at skin incision
  Arms: saline-lidocaine-morphine (SLM)

SUMMARY:
Epidural chloroprocaine is often used in obstetrical anesthesia because of its fast onset and short duration. These properties make it an ideal drug to use for epidural anesthesia in patients undergoing postpartum tubal ligation. When epidural morphine is given after chloroprocaine, there is a decreased efficacy of analgesia as compared to lidocaine (1). Several studies have hypothesized a specific opioid receptor mediated antagonism of chloroprocaine (2,3). Karambelkar raised the question whether this decreased efficacy is due to a disparity between the time the chloroprocaine anesthesia resolves and the onset of epidural morphine analgesia, resulting in a time window of pain (2). The duration of action of epidural 2-CP anesthesia is 30-45 minutes and the onset of epidural morphine analgesia is 60-70 minutes, therefore the regression of sensory blockade before the onset of the morphine analgesia could result in a window of pain (2). Hess and colleagues studied epidural morphine analgesia and women who had a Cesarean delivery under spinal bupivacaine anesthesia (3). Subjects were randomized to receive epidural 2-CP and morphine or epidural saline and morphine. There was no difference in postoperative analgesia between the two groups (3 and personal communication, Dr. Philip Hess). A literature search cross referencing epidural chloroprocaine, using Pub Med, did not produce any articles comparing epidural morphine given before the procedure (in an attempt to time the onset of analgesia with the resolution of chloroprocaine anesthesia) to the standard administration time after the procedure.

DETAILED DESCRIPTION:
Women undergoing post partum tubal ligation with an epidural in-situ will be randomly double blindedly selected into one of three groups for pain control. The groups are epidural 1) epidural morphine-chloroprocaine 2) epidural chloroprocaine-morphine 3) epidural morphine-lidocaine. Groups 1 and 3 will receive morphine 30 minutes prior to local anesthetic dosing followed by saline placebo after local dosing. Group 2 will receive placebo 30 minutes prior to local anesthetic dosing followed by epidural morphine. Pain scores and supplemental analgesic requirements will be evaluated 30 minutes, 1hr, 2hr, 4hr and every 4 hrs for the first 24hrs.

ELIGIBILITY:
Inclusion Criteria:

* All patients with an epidural catheter in situ for labor analgesia, status post a vaginal delivery, and scheduled for a postpartum tubal ligation under epidural anesthesia will be eligible

Exclusion Criteria:

* Allergy/hypersensitivity to morphine
* Allergy/hypersensitivity to ester-linked local anesthetics or para-amino benzoic acid (PABA)
* Body Mass Index >40 kg/m2
* Patients using chronic opioids
* History of obstructive sleep apnea
* Any contraindication to epidural anesthesia

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2004-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Wong, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Eisenach JC, Schlairet TJ, Dobson CE 2nd, Hood DH. Effect of prior anesthetic solution on epidural morphine analgesia. Anesth Analg. 1991 Aug;73(2):119-23. doi: 10.1213/00000539-199108000-00003. PMID 1854026
- [Background] Karambelkar DJ, Ramanathan S. 2-Chloroprocaine antagonism of epidural morphine analgesia. Acta Anaesthesiol Scand. 1997 Jun;41(6):774-8. doi: 10.1111/j.1399-6576.1997.tb04782.x. PMID 9241341
- [Background] Camann WR, Hartigan PM, Gilbertson LI, Johnson MD, Datta S. Chloroprocaine antagonism of epidural opioid analgesia: a receptor-specific phenomenon? Anesthesiology. 1990 Nov;73(5):860-3. doi: 10.1097/00000542-199011000-00011. PMID 2173443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 136 subjects approached and assessed for eligibility
Pre-assignment Details: Excluded from randomization (n=37), 26 refused to participate, 11 did not meet exclusion criteria
Groups:
- Morphine - 2 Chloroprocaine - Saline (MCS): morphine will be administered 30 min prior to epidural anesthesia; 2CP will be used to achieve a T4 level; saline will be administered at skin incision
- Saline-2 Chloroprocaine - Morphine (SCM): saline will be administered 30 min prior to epidural anesthesia; 2-chloroprocaine will be used to achieve a T4 level; morphine will be administered at skin incision
- Saline - Lidocaine - Morphine (SLM): Saline administered 30 minutes prior to lidocaine to achieve a T4 anesthesia level. Morphine administered at skin incision.
Period: Overall Study
Arm/Group | Morphine - 2 Chloroprocaine - Saline (MCS) | Saline-2 Chloroprocaine - Morphine (SCM) | Saline - Lidocaine - Morphine (SLM)
Started | 33 | 33 | 33
Completed | 29 | 30 | 28
Not Completed | 4 | 3 | 5
Not completed — Did not receive intervention | 4 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine - 2 Chloroprocaine - Saline (MCS) | Saline-2 Chloroprocaine - Morphine (SCM) | Saline - Lidocaine - Morphine (SLM) | Total
Number analyzed (Participants) | 33 | 33 | 33 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 33 | 33 | 99
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (4) | 31 (5) | 29 (4) | 30 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 33 | 99
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 33 | 99

OUTCOME MEASURES:

1. Primary Outcome: Duration of Continuing Analgesia
Description: Time to first request for supplemental analgesia
Time Frame: 48 hours
Population: All participants receiving the intervention were analyzed
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Morphine - 2 Chloroprocaine - Saline (MCS) | Saline-2 Chloroprocaine - Morphine (SCM) | Saline - Lidocaine - Morphine (SLM)
Number analyzed (Participants) | 29 | 30 | 28
hours | 28.6 [4.4 to 52.7] | 2.2 [0 to 4.8] | 25.8 [10.7 to 40.9]
Statistical Analysis 1: Comparison: Morphine - 2 Chloroprocaine - Saline (MCS); A sample of 56 was estimated to have an 80% power to detect a 30% difference in the proportion of subjects with continuing analgesia in the MCS versus the SCM groups when 50% of the subjects in the SCM had requested supplemental analgesia. 28 subjects was added to compare the influence of time of morphine and 2-chloroprocaine administration to lidocaine-morphine analgesia. The primary outcome was compared using Kaplan-Meier survival analysis and the log-rank test; Test type: Superiority or Other; p = 0.006, Log Rank
Statistical Analysis 2: Comparison: Morphine - 2 Chloroprocaine - Saline (MCS) vs Saline-2 Chloroprocaine - Morphine (SCM); Test type: Superiority or Other; p = 0.83, Log Rank
Statistical Analysis 3: Comparison: Saline-2 Chloroprocaine - Morphine (SCM); Test type: Superiority or Other; p = 0.009, Log Rank

2. Secondary Outcome: Verbal Rating Score (0 to 10) for Pain (VRPS)
Description: Verbal Rating Pain Score (VRPS) at time of post-anesthesia recovery room entry, where 0 = no pain and 10 = worst pain imaginable
Time Frame: At recovery room entry
Population: Verbal Rating Score for Pain (0-10) where 0 = no pain and 10 = worst pain imaginable
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Morphine - 2 Chloroprocaine - Saline (MCS) | Saline-2 Chloroprocaine - Morphine (SCM) | Saline - Lidocaine - Morphine (SLM)
Number analyzed (Participants) | 29 | 30 | 28
Scores on a scale | 2 [0 to 4.5] | 2 [1.8 to 4.0] | 0 [0 to 1.5]
Statistical Analysis 1: Comparison: Morphine - 2 Chloroprocaine - Saline (MCS) vs Saline - Lidocaine - Morphine (SLM); Test type: Superiority or Other; p < 0.05, Kruskal-Wallis
Statistical Analysis 2: Comparison: Saline-2 Chloroprocaine - Morphine (SCM) vs Saline - Lidocaine - Morphine (SLM); Test type: Superiority or Other; p < 0.05, Kruskal-Wallis

3. Primary Outcome: Supplemental Analgesia in First 90 Minutes
Description: Participants requesting supplemental analgesia in the first 90 minutes following study drug
Time Frame: 90 min
Measure: Number; unit: participants
Arm/Group | Morphine - 2 Chloroprocaine - Saline (MCS) | Saline-2 Chloroprocaine - Morphine (SCM) | Saline - Lidocaine - Morphine (SLM)
Number analyzed (Participants) | 29 | 30 | 28
participants | 0 | 10 | 0
Statistical Analysis 1: Comparison: Morphine - 2 Chloroprocaine - Saline (MCS) vs Saline-2 Chloroprocaine - Morphine (SCM); Test type: Superiority or Other; p = 0.01, Chi-squared, Corrected
Statistical Analysis 2: Comparison: Saline-2 Chloroprocaine - Morphine (SCM) vs Saline - Lidocaine - Morphine (SLM); Test type: Superiority or Other; p = 0.01, Chi-squared, Corrected

4. Secondary Outcome: Supplemental Analgesia in First 48 Hours
Description: Participants requesting supplemental analgesia in first 48 hours
Time Frame: 48 hours
Measure: Number; unit: Participants
Arm/Group | Morphine - 2 Chloroprocaine - Saline (MCS) | Saline-2 Chloroprocaine - Morphine (SCM) | Saline - Lidocaine - Morphine (SLM)
Number analyzed (Participants) | 29 | 30 | 28
Participants | 12 | 8 | 12
Statistical Analysis 1: Comparison: Morphine - 2 Chloroprocaine - Saline (MCS) vs Saline-2 Chloroprocaine - Morphine (SCM); Test type: Superiority or Other; p = 0.20, Chi-squared, Corrected

ADVERSE EVENTS:
Arm/Group | Morphine - 2 Chloroprocaine - Saline (MCS) | Saline-2 Chloroprocaine - Morphine (SCM) | Saline - Lidocaine - Morphine (SLM)
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/28

LIMITATIONS AND CAVEATS:
We used a single 30-minute interval between morphine and 2-chloroprocaine administration and additional investigation is warranted to determine the optimum interval for administration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No